CLINICAL TRIAL: NCT06704399
Title: Investigation of the Effect of Acceptance and Commitment Therapy-Based Psychoeducation on Rumination and Self-Compassion in Patients Diagnosed With Panic Disorder: Randomized Controlled Study
Brief Title: Psychoeducation Based on Acceptance and Commitment Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatmanur ÖZCAN MİRCALI, Principal investigator, PhD student, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MuglaSKU-HEM-FOM-01
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Panic Disorder
Keywords: rumination; self-compassion
MeSH Terms: conditions — Panic Disorder; Rumination Syndrome | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Two groups included experimental and control group, pre-test, post-test and follow-up test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- psycoeducation (Active Comparator): Psychoeducation based on acceptance and commitment therapy will be applied to the experimental group of 25 people. Pre-test, post-test and follow-up test will be applied.
  Interventions: Other: Acceptance and Commitment Therapy-Based Psychoeducation
- control (Active Comparator): No intervention will be applied to the control group of 25 people. Pre-test, post-test and follow-up test will be applied.

INTERVENTIONS:
Other: Acceptance and Commitment Therapy-Based Psychoeducation — Psychoeducation based on acceptance and commitment therapy will be applied to the experimental group.
  Arms: psycoeducation
Other: control group — No intervention will be applied to the control group.

SUMMARY:
The aim of this study is to manage individual psychoeducation in acceptance and commitment therapy for problems with panic disorder and to evaluate the effect of this program on rumination and self-resilience.

DETAILED DESCRIPTION:
Panic disorder; palpitations, sweating, tachycardia, fear of death, depersonalization, derealization, fear of going crazy, etc. It is a psychiatric disorder with symptoms. The most commonly used psychotherapy method for panic disorder patients is cognitive behavioral therapies. Acceptance and Commitment Therapy is a psychotherapy method originating from cognitive behavioral therapy. Acceptance and Commitment Therapy helps individuals act in the direction of their values by allowing them to contact their painful experiences rather than trying to escape or try to get rid of their difficult experiences, thoughts, and feelings. Acceptance and Commitment Therapy supports psychological well-being by providing psychological flexibility in the person. Rumination is mental rumination, which is used to keep thoughts spinning in the mind repetitively after an event.Self-compassion is a concept used to mean understanding oneself despite one's mistakes. This study aims to create psychoeducation based on acceptance and commitment therapy for patients with panic disorder and to evaluate the effect of this program on rumination and self-compassion. Psychoeducation, an evidence-based practice, is very important for the nursing profession. Although nurses have a significant impact on psychoeducational practices, this role is ignored and not implemented adequately. In addition, since there is no research examining the concepts of rumination and self-compassion together in people with panic disorder, it is thought that our study will be useful in new research.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Panic Disorder followed in Muğla Training and
* Research Hospital Psychiatry Polyclinics,
* Those between the ages of 18-65 who agree to participate in the research,
* Those who were in a euthymic mood during the interview, according to physician control,
* Those who speak Turkish,
* Those who are literate,
* Those who have a computer and internet access for the program to be conducted online if deemed necessary during the research process,
* Not having undergone such training within the last year is within the scope of the inclusion criteria.

Exclusion Criteria:

* Having a diagnosis of a psychiatric disease in addition to panic disorder,
* Having an attack period during the training period,
* Individuals with cognitive (diagnosed by a physician) and physical disability (hearing, speaking, etc.) are included in the exclusion criteria from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Ruminative Thought Style Questionnaire | 7 week
  The scale is a 7-point Likert type consisting of 20 items. 7 = Very good and 1 = Not at all, and participants are asked to score each item according to how much it reflects themselves. The internal consistency coefficient of the scale, Cronbach's alpha value, was found to be .907. In the item analysis, the item total score correlation was calculated and the total correlations of the items were found to be between 0.474 and 0.699.

SECONDARY OUTCOMES:
Self Compassion Scale | 7 week
  The original Self-Compassion Scale consists of 6 subscales containing 26 items. The scale is a 5-point Likert type and those who answer "almost never = 1 and almost always = 5" are asked to rate how often they move. The Turkish form of the self-compassion scale, unlike the original, consists of 24 items because the scale shows a unidimensional structure and at the same time, 2 items with item-total correlations below 30 were removed from the scale. The internal consistency coefficient of the scale was calculated as .89 and the test-retest correlation was calculated as .83.

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Sıtkı Koçman University, Muğla, mentese, Turkey (Türkiye)